CLINICAL TRIAL: NCT05017493
Title: Treatment of Early-Stage Covid-19 With a Herbal Compound, Xagrotin
Brief Title: Treatment of Covid-19 With a Herbal Compound, Xagrotin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biomad AS (Industry)
Collaborators: Directorate of Health of Sulaimani, Iraq (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-032021-SULXAG/NO
Record Dates: First submitted 2021-04-04; First posted 2021-08-24 (Actual); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Patients in the Treatment arm received Xagrotin in combination to the standard of care for Covid19.
  Interventions: Combination Product: Xagrotin
- Control arm (No Intervention): Patients in the Control arm received the standard of care for Covid19.

INTERVENTIONS:
Combination Product: Xagrotin — A group of patients were treated with Xagrotin with or without standard of care, the control group received stadard of care
  Arms: Treatment arm

SUMMARY:
This is an interventional, multi-center, randomized study. Adults with confirmed covid-19 disease not more than 10 days before enrollment date were recruited (n=361). Patients in same condition who had treated with standard of care were randomly assigned to the control group (n=178). The investigators analyzed the effect of a herbal compound, Xagrotin, and also investigated impact of different characteristics for instance gender, age, duration of disease, smoking habits and concomitant diseases on the outcome.

DETAILED DESCRIPTION:
This is an interventional, multi-center, randomized study that has been performed in an outpatient setting (n=361). Adults with confirmed covid-19 disease not more than 10 days before enrollment date were recruited. Patients in same condition who had treated with standard of care were randomly assigned to the control group (n=178). The investigators analyzed the effect of a herbal compound, Xagrotin, and also investigated impact of different characteristics for instance gender, age, duration of disease, smoking habits and concomitant diseases on the outcome. Adverse events were registered.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or higher
* Newly diagnosed (no longer than 10 days)
* PCR or clinically confirmed Covid-19

Exclusion Criteria:

* Severe pulmonary disease
* Severe cardiovascular disease
* Severe hepatic disease
* Severe renal disease
* Diabetes mellitus type one
* Metabolic acidosis
* Oxygen saturation <70%
* Pregnancy
* Breast feeding
* Concomitant treatment with anticoagulation drugs
* Concomitant treatment with CYP3A4 medicines with narrow therapeutic window

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2021-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Directorate of health of Sulaimani, Iraq -KRG, Sulaymaniyah, Iraq

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All adult patients in an outpatient setting who were confirmed as coronavirus patients were eligible to be included in the study.
Pre-assignment Details: Age 18 or higher, Newly diagnosed (no longer than 10 days), PCR or clinically confirmed Covid-19
Period: Overall Study
Arm/Group | Treatment Arm | Control Arm
Started (483 patients enrolled in treatment arm) | 483 | 178
Treatment & Care (483 patients received Xagrotin) | 483 | 178
Follow up (483 patients were followed up) | 483 | 178
Mortality Check (483 patients were checked for mortality) | 483 | 178
Completed (361 patients completed pr protocol) | 361 | 178
Not Completed | 122 | 0
Not completed — Withdrawal by Subject | 26 | 0
Not completed — Physician Decision | 15 | 0
Not completed — Protocol Violation | 81 | 0

BASELINE CHARACTERISTICS:
Population: Both paitients who received and NOT received Xagrotin
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Control Arm | Total
Number analyzed (Participants) | 483 | 178 | 661
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 5 | 28
  Between 18 and 65 years | 397 | 150 | 547
  >=65 years | 63 | 23 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (17.16) | 44.297 (17.16) | 44.1 (17.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 91 | 303
  Male | 271 | 87 | 358
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 483 | 178 | 661
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Iraq | 483 | 178 | 661

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Number of Participants who died by day 30 after the enrollment
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 361 | 178
participants | 2 | 10

2. Secondary Outcome: Duration of Disease From Beginning of Treatment
Description: Number of days the patient has experienced the symptoms
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 361 | 178
Days | 9.9 (5.5) | 18.1 (9.5)

3. Secondary Outcome: Hospitalization
Description: Number of participants who have been hospitalized for Covid-19
Time Frame: 30 days
Measure: Number; unit: Participatnts
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 361 | 178
Participatnts | 11 | 57

4. Secondary Outcome: Duration of Hospitalization When Occurred
Description: Days the participants were hospitalized
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 361 | 178
Days | 5.56 (4.94) | 5.5 (3.42)

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | Treatment Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 2/483 | 10/178
Serious Adverse Events (participants affected / at risk) | 1/483 | 10/178
Other Adverse Events (participants affected / at risk) | 113/483 | 15/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=483) | Control Arm (N=178)
Xagrotin (Blood and lymphatic system disorders) | 1 (1) | 10 (10) — Xagrotin is a herbal compound, and it contains flavonoids, phenols, etc., which dilate blood vessels. Therefore, the risk of internal bleeding is higher in people who take high-dose vasodilators and high-dose Xagrotin at the same time.
OTHER ADVERSE EVENTS (reported when occurring in more than 2.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=483) | Control Arm (N=178)
Diarrhea (Gastrointestinal disorders) | 113 (113) | 15 (15) — Participants got Diarrhea
Flatulence (Gastrointestinal disorders) | 113 (113) | 15 (15) — Participants got flatulence

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs discuss or publish the results only according to a prior agreement with the sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT05017493/Prot_003.pdf
  • Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT05017493/SAP_004.pdf